CLINICAL TRIAL: NCT06753357
Title: Prevalence of Cancer Rehabilitation Needs and Drivers of Rehabilitation Service Uptake in Breast Cancer Survivors
Brief Title: Breast Cancer Rehabilitation Needs and Service Uptake
Status: Not yet recruiting | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RIG202403-006PR
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Cancer Survivorship; Health Attitude
Keywords: Breast cancer; Cancer rehabilitation; Rehabilitation needs; Rehabilitation service uptake; Cancer survivorship; Health Belief Model; Technological enablers
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Eligible patients: Female patients from the Breast Surgery clinic at Changi General Hospital (with referrals from the on-site Medical Oncology clinic). A consecutive purposive sample of 400 participants will be recruited. There are no race-based or minority-based subject restrictions. Male patients with breast cancer are rare and are thus excluded from recruitment. Patients will be approached by a clinical research co-ordinator (CRC) or study team member who will explain the study and seek consent for recruitment.

SUMMARY:
The investigators are attempting to verify the prevalence of cancer rehabilitation needs at our institution in breast cancer patients. The investigators also want to assess 1) self-perceived needs for cancer rehabilitation services, 2) awareness, willingness, and patient health beliefs as determinants for cancer rehabilitation-seeking behaviour, and 3) the modifiable patient factors driving the mismatch between needs and uptake in our population.

Patients attending outpatient clinics in our hospital will be approached to answer a questionnaire designed to find out this information. The investigators hope that the results will ultimately inform the design of better triage and referral systems that match patients to services based on their rehabilitation needs.

The investigators believe that local survivors of breast cancer have unmet rehabilitation needs and that it is possible to evaluate their readiness to seek access to rehabilitation services as well as identify mismatches between provided and desired services through the administration of a cancer rehabilitation questionnaire (CRQ).

DETAILED DESCRIPTION:
STUDY DESIGN The study is conceptualised as a cross-sectional observational study of breast cancer survivors in a multiethnic urban Asian population that is representative of our demographic. It will conform to the STROBE guidelines. The study will be registered prior to site initiation. Ethics approval is pending.

STUDY POPULATION Consecutive purposive sample of all female patients with breast cancer in the Breast Surgery clinics (with Medical Oncology as a referring site).

CONDUCT OF STUDY The study will take place in the specialist outpatient clinics in CGH. All unique patients attending their clinic appointments will be screened. Patients fulfilling the inclusion and exclusion criteria will be approached for recruitment and enrolment. They will complete the questionnaire and provide relevant demographic features in the same sitting, within a private room. Verbal translation into Mandarin, Malay, or Tamil by the administrator will be done for patients who are unable to communicate in English. No audio or video recording will be performed.

CANCER REHABILITATION QUIESTIONNAIRE (EXPANDED) The Cancer Rehabilitation Questionnaire (CRQ) was designed by a team at the National University Hospital, Singapore, to investigate the functional problems faced by cancer survivors as well as their attitudes toward participation in rehabilitation. It comprises 12 common cancer-associated functional issues with yes/no answers, as well as further qualitative questions to explore barriers to participation in rehabilitation. The original tool was validated, with strong internal consistency and had a large effect size for differentiating clinically-significant declines in physical functioning. However, it was administered a decade ago and not optimised specifically for contemporary patients with breast cancer.

The investigators evaluated the components of the CRQ based on suitable available literature, and have expanded it with 2 more parts to reflect the increasing role of technology in healthcare delivery, allow patients to open-endedly discuss desired rehabilitation and therapy services, as well as explore concerns and health-seeking behaviours specific to breast cancer impairments and post-treatment sequelae.

1. The first part (Expanded Questions) includes additional symptoms and impairments that are specific to breast cancer survivors such as changes in appearance, hot flashes, and mood lability. Along with symptoms and impairments from the original CRQ, patients will be asked to grade their symptoms by severity, as well as judge the kind of rehabilitative service they will need, if any (ranging from information leaflets and community-based rehabilitation to specialised medical evaluation and clearance). It also includes service-specific questions relating to the need for prehabilitation as well as acceptability of telerehabilitation, which is becoming a relevant treatment model in the post-COVID-19 environment. Questions are based on previously-uncovered barriers. A single open-ended question will seek feedback on lacking services as perceived by patients.
2. The second part (Health Beliefs) includes 29 questions based on factors causing patients to not utilise cancer rehabilitation services, based on previous focus group work in older breast cancer survivors in the USA, and designed based on the HBM and healthcare-related studies that have utilised it. Questions examine patients' perceived susceptibility to worse health state owing to their cancer and its treatment (4 questions), their assessment of its severity on their lifestyle (4 questions), perceived benefits of participating in cancer rehabilitation (4 questions), and any barriers that would impede them from accessing cancer rehabilitation services (10 questions). Additional questions for likelihood of health behaviour examine their self-efficacy in successfully carrying out behaviour change (3 questions) as well as responsiveness to potential cues to taking action (3 questions). Responses are rated on a five-point Likert scale.
3. A final section requires capture of the patients' back-end data such as treatment status, treatment type, comorbidities, and rehabilitation needs triage based on the physician's assessment of their needs. It will be validated against patients' self-assessments as well as contemporary work.

STATISTICAL AND ANALYTIICAL PLANS Descriptive statistics of patient demographic and clinical characteristics will be reported as number and percent for categorical data, mean ± standard deviation (SD) for normally distributed data, and median and interquartile range (IQR) for non-normally distributed data. The prevalence of reported symptoms and impairments will be reported as number and percent of patients, with the corresponding 95% confidence intervals (CIs) of the population percentages.

Multivariable linear regression will be used to assess if reported impairments and impairment severity are independently associated with patients' self-assessed need for rehabilitative services. The linearity assumption will be assessed using the Box-Tidwell test, the homoscedasticity assumption using a plot of model residuals against fitted values, and the normality assumption using a quantile-quantile (Q-Q) plot. Cohen's Kappa (κ) will be used to examine agreement between patients' self-assessed need for rehabilitation and level of care needed, against physician-assessed needs and level of care required, as they are categorical variables.

Results for the questions pertaining to technology-enabled rehabilitation and barriers to rehabilitation will be reported through central tendency measures (mean ± SD or median + IQR, with 95% CIs). This is likewise for the Likert-type items that make up the Health Beliefs construct. Internal consistency of the health belief questions that evaluate the same concept will be assessed using Cronbach's alpha. Data will be tabulated and analysed using IBM SPSS Statistics version 26.0 (IBM Corp, Armonk, NY, USA). No interim analysis is necessary as the study is not conceptualised as a randomised controlled trial.

WITHDRAWAL FROM THE STUDY Subjects may withdraw voluntarily from participation in the study at any time, including after completion, with no prejudice to their clinical care or outpatient follow-up. Their data will be removed from the electronic records, and the hardcopy data collection form will be physically destroyed. Their withdrawal will be reported in the STROBE flowchart subsequently.

DISCONTINUATION OF THE STUDY The study may be discontinued for any of the following reasons.

1. Adverse event or serious adverse event related to data collection or study conduct, which implicates safety of subsequent recruits
2. Other unforeseen circumstances In the event of study discontinuation, the investigators will inform the CIRB accordingly and the study team will evaluate the incomplete data to determine if there is sufficient scholarly merit remaining to justify write-up and publication.

SAFETY MONITORING PLAN Patients will be under the care of a trained study team member or CRC during recruitment and questionnaire administration. They will be monitored for discomfort during this period. Other clinical deteriorations will be managed routinely. Data will be reviewed on a monthly basis by an appointed co-investigator for integrity as well as completion. This includes screening and recruitment figures, as well as demographics, functional/clinical characteristics, as well as questionnaire responses. Data safety will be through lock-and-key storage of physical documents as well as access-restricted, password-protection for electronic data, which can only be viewed on the hospital's intranet-facing devices.

DATA ENTRY AND STORAGE Demographic data will be collected from patients' electronic medical records. Anthropometric and clinical measurements will be collected physically. All records will be recorded in a hardcopy data collection form to be filed in the Investigator Site File (ISF) that is stored under lock-and-key in the Research Office. All data will be transcribed electronically into REDCap which is hosted on the hospital's intranet and is access-restricted as well as password-protected. Only study team members (including the clinical research co-ordinator) will have access to the data. Data will be de-identified prior to analysis by the statistician. All data will be kept for 7 years post-completion or post-publication, whichever is later. Following that, electronic data will be deleted and all paper records will be physically destroyed.

DATA QUALITY ASSURANCE All data will be collected by a small pre-defined group of trained medical doctors and clinical research co-ordinators with medical backgrounds. All study team members will be pre-trained and briefed on the administration of the questionnaire. All data will be collected during the questionnaire administration, except for the Charlson Comorbidity Index which will require access to the patient's Electronic Medical Records (EMR). All study team members will have previous training and experience in accessing the patients' EMR.

ETHICAL CONSIDERATIONS This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and that are consistent with the Good Clinical Practice and the applicable regulatory requirements. The principal investigator is responsible for informing the CIRB of any amendments to the protocol or other study-related documents, as per local requirement.

INFORMED CONSENT Informed consent will be collected prior to administration of a questionnaire. Patients will be screened upon registration in the respective clinics. Eligible patients would then be approached for consent while they are on-site. All study team members would be trained and hence eligible for consent-taking. Consent will be taken physically and in writing. Risks and benefits of participation will be clearly explained. Patients will be given ample time to make a decision and/or decline with no impact on their standard of clinical care. If a family member's presence is requested or deemed necessary but they cannot be present in the premises, the patient will not be recruited in that instance. The investigators will not consider remote consent as our target demographic is generally ambulant.

The requirement for a witness for all consent-taking is exempted as the study comprises solely of a survey under Regulation 26 of the Human Biomedical Research Regulations 2017 (not invasive, not interventional, not restricted human biomedical research). A legally-authorised representative (LAR) would not be required. Upon enrolment into the study, a note will be entered into the patient's electronic medical record. For non-English speakers, the investigators will use appropriate translation (in Mandarin, Malay, or Tamil) performed by the study team member or CRC. Patients with cognitive impairment meeting the diagnostic criteria for major neurocognitive disorder will not be recruited as this may affect the accuracy of their answers. The study team member assessing for cognitive impairment would have been satisfactorily trained prior. They will be treated as a vulnerable population and excluded from recruitment.

The investigators do not foresee the recruitment of other special populations such as children, prisoners, or other vulnerable individuals. In obtaining and documenting informed consent, the investigator should comply with the GCP guidelines and to the ethical principles that have their origin in the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Age 21yrs old and above
3. Histological diagnosis of breast cancer at any stage (or clinical consensus at a Tumour Board meeting, for example if the condition is metastatic and biopsy is not indicated for any reason)
4. Started treatment (surgical, medical, radiotherapeutic, or otherwise) with curative or palliative intent
5. Speak English, Mandarin, or Malay, or Tamil, and are able to understand a verbally-translated version of the questionnaire
6. Able to provide informed consent

Exclusion Criteria:

1. Unable to answer the questionnaire for any reasons such as cognitive impairment or sensory dysfunction
2. Declined participation

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive purposive sample of all female patients with breast cancer in the Breast Surgery and Medical Oncology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Symptom/impairment prevalence | At the point of recruitment
  The prevalence of reported symptoms and impairments among breast cancer survivors.

SECONDARY OUTCOMES:
Awareness of available support | At the point of recruitment
  Awareness of available support for symptomatic patients
Willingness to receive support | At the point of recruitment
  Willingness to receive rehabilitation support for symptomatic patients
Health beliefs in relation to receiving rehabilitation support | At the point of recruitment
  Factors associated with the uptake of such sessions (using the HBM factors as well as sociodemographic factors of age, treatment status, social support, and highest education level)
Agreement on level of care | At the point of recruitment
  Agreement between patient and physician for the level of care they feel would be appropriate for their case (unsupervised exercise, supervised community-based rehabilitation, clinically-supervised rehabilitation, rehabilitation medicine consult, or exercise clearance/work-up). The professional judgement will be from a rehabilitation medicine physician with experience managing patients with cancer rehabilitation needs.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund JR Neo, MBBS MRCP, Principal Investigator — Singapore Health Services Pte Ltd
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Data is protected under the SingHealth Data Protection Policy which is compliant to the Singapore Personal Data Protection Act 2012